CLINICAL TRIAL: NCT03885219
Title: Prospective Phase II Single-arm Study of Nab-paclitaxel and S-1 in Patients With Locally Advanced Pancreatic Cancer.
Brief Title: Nab-paclitaxel and S-1 in Patients With Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-1751
Record Dates: First submitted 2019-02-20; First posted 2019-03-21 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nab-paclitaxel and S-1 (Experimental): chemotherapy of Nab-Paclitaxel and S-1, repeat 21 days for up to 8 cycles. The following treatment including pancreatectomy, continuing same chemotherapy, S-1 maintenance therapy, or radiotherapy will be decided after discussion between physicians and patients.
  Interventions: Drug: Nab-paclitaxel and S-1

INTERVENTIONS:
Drug: Nab-paclitaxel and S-1 — Nab-paclitaxel: 120 mg/m2 d1, 8, S-1:Body surface area < 1.25 m2, 80 mg/d; Body surface area ≥ 1.25 m2 , < 1.5 m2, 100 mg/d; Body surface area ≥1.5 m2, 120 mg/d; Bid, d1-14; repeat every 21 days.

SUMMARY:
This study is a single-arm, multi-center, open-label prospective phase II clinical study designed to evaluate the efficacy and safety of nab-paclitaxel and S-1 in patients with locally advanced pancreatic cancer. A total of 60 subjects who meet the criteria will be treated with nab-paclitaxel and S-1. The primary endpoint is 6 months progression free survival rate, and secondary endpoints include objective response rate, overall survival, progression free survival and toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have good compliance, can understand the research process of this study, and sign a written informed consent
2. Patients with pathologically confirmed pancreatic adenocarcinoma.
3. Patients who have not received prior chemotherapy, radiotherapy or other systematic treatment for pancreatic cancer;
4. Patients with locally advanced pancreatic cancer ( NCCN Version 1，2019 criteria).
5. ECOG PS 0-1;
6. Tumor size is measurable according to RECIST1.1 criteria
7. Expected survival over 3 months;
8. Bone marrow function: neutrophils≥1.5x109/L, platelets ≥100x109/L, hemoglobin≥ 90g/L;
9. Liver and kidney function: serum creatinine≤1.5ULT; AST and ALT≤ 2.5 ULT; total bilirubin ≤ 1.5 ULT;
10. No contraindications to the use of S-1 and nab-paclitaxel.

Exclusion Criteria:

1. ≥ Grade 2 existing peripheral neuropathy;
2. Any other malignancy within 5 years prior to enrollment, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, bladder, or nonmelanomatous skin cancer.
3. Active, uncontrolled infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate treatment.
4. Severe, active co-morbidity, defined as follows:

   Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months Transmural myocardial infarction within the 6 months of study registration Uncontrolled hypertension, diabetes or arrhythmia. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization.
5. Not able to take medicine orally.
6. Pregnancy or lactation, and women of childbearing age who refused to take appropriate contraceptive measures during the course of this study;
7. Participation in other clinical trial within 30 days before the first dose of the drug;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival (PFS) | 6 months
  The proportion of patients who did not experience disease progression or die from disease progression within 6 months from the registration.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  Refers to the proportion of patients with partial tumor remission (PR) and complete remission (CR).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided